CLINICAL TRIAL: NCT01941485
Title: A Prospective, Global, Multi-Center Study to Evaluate Longitudinal Flap Accuracy on Subjects Undergoing Myopic Refractive Surgery Using the WaveLight® Refractive Suite
Brief Title: WaveLight® Refractive Flap Accuracy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A01354
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Refractive Error
Keywords: nearsighted; astigmatism; LASIK; refractive surgery; WaveLight
MeSH Terms: conditions — Refractive Errors; Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WaveLight Refractive Suite (Experimental): LASIK surgery (laser in situ keratomileusis) per standard of care
  Interventions: Device: WaveLight® Refractive Suite; Procedure: LASIK surgery

INTERVENTIONS:
Device: WaveLight® Refractive Suite — Excimer EX500 and Femtosecond FS200 lasers (Wavelight® Refractive Suite) used during LASIK surgery for corneal flap creation and corneal ablation
Procedure: LASIK surgery — Surgical procedure for treating refractive error based on corneal reshaping

SUMMARY:
The purpose of this study is to evaluate the accuracy of the WaveLight FS200 femtosecond laser, as assessed by 1 day and 1 month post-operative optical coherence tomography (OCT) anterior segment corneal measurements compared to pre-operative flap thickness target.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign an informed consent form.
* Have refractive error (in both eyes) that requires refractive surgery.
* Willing to undergo LASIK surgery using the Wavelight® Refractive Suite.
* Myopia between 0.00 to -12.0 Diopters pre-operatively.
* Astigmatism between 0.00 to +6.00 Diopters pre-operatively.
* Willing and able to attend post-operative examinations per protocol schedule.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Participation in a clinical study within the last 30 days.
* History of previous corneal surgery in either eye.
* Multifocal ablations in either eye.
* PRK or PTK surgery in either eye.
* Suffering from acute or recurring eye diseases in either eye, such as corneal ulcers, cataract, etc.
* Any ocular disease and/or condition that, in the Investigator's clinical judgment, may put subject at significant risk, compromise study results, or interfere significantly with subject's participation in the study.
* Unable to discontinue contact lens wear as specified in protocol.
* History of Herpes simplex or Herpes zoster keratitis.
* Active ocular rosacea.
* Lyme disease.
* Severe ocular allergies.
* Other medical conditions and use of medications as specified in protocol.
* Pregnant or planning to become pregnant during the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, GCRA, Global Med Affairs, Operations, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in the US and 1 study center located in Greece.
Pre-assignment Details: Of the 60 enrolled subjects, 1 was exited as a screen failure prior to surgery. This reporting group includes all enrolled subjects who underwent LASIK surgery (59).
Groups:
- WaveLight Refractive Suite: Excimer EX500 and Femtosecond FS200 lasers used during LASIK surgery for corneal flap creation and corneal ablation
Period: Overall Study
Arm/Group | WaveLight Refractive Suite
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled subjects who underwent LASIK surgery (59).
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (9.22)
Gender [Count of Participants; unit: Participants]
  Female | 34
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between Achieved Flap Thickness at Day 1 Postoperative as Assessed by OCT and Expected Flap Thickness as Determined Pre-operatively
Description: The expected flap thickness as determined pre-operatively was subtracted from the achieved flap thickness at Day 1 postoperative as assessed by optical coherence tomography (ie, an imaging method using light to capture three-dimensional images). Accuracy of flap creation was defined as an achieved thickness within 10 microns of expected thickness.
Time Frame: Day 1 Postoperative
Population: This analysis population includes all subjects with 1 day post-operation measurements of the primary effectiveness endpoint.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 59
microns
  Right eye (OD) | 14.996 (12.7509)
  Left eye (OS) | 13.644 (10.4762)

2. Secondary Outcome: Incidence of Development of Opaque Bubble Layer (OBL)
Description: OBL (the collection of gas bubbles during corneal flap creation) was assessed by digital photo analysis of the area covered by the flap and is reported as the percentage of participants with opaque bubble layer development during femtosecond flap creation.
Time Frame: Operation/Surgery (Day 1)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 59
percentage of participants
  Right eye (OD) | 20.3
  Left eye (OS) | 35.6

3. Secondary Outcome: Extent of Opaque Bubble Layer (OBL) Within the Femtosecond Flap
Description: The extent of OBL was assessed by digital photo analysis of the area covered by the flap and is reported as the percentage of flap with opaque bubble layer development during femtosecond flap creation.
Time Frame: Operation/Surgery (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of flap
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 59
percentage of flap
  Right eye (OD) | 8.9 (7.59)
  Left eye (OS) | 11.1 (6.94)

4. Secondary Outcome: The Difference Between Achieved Flap Thickness at Month 1 Post-operative as Assessed by OCT and Expected Flap Thickness as Determined Preoperatively
Description: The expected flap thickness as determined pre-operatively subtracted from the achieved flap thickness at Month 1 postoperative as assessed by optical coherence tomography (ie, an imaging method using light to capture three-dimensional images). Accuracy of flap creation was defined as an achieved thickness within 10 microns of expected thickness.
Time Frame: Month 1 Postoperative
Population: This analysis population includes all subjects with 1 month post-operative measurements of the primary efficacy endpoint with data at the specific time point.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 58
microns
  Right eye (OD) | 8.638 (5.5177)
  Left eye (OS) | 8.207 (4.7564)

5. Secondary Outcome: Uncorrected Visual Acuity (UCVA)
Description: Visual acuity (VA) without spectacles or other visual corrective devices, was performed with an Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at a distance of 4 meters. UCVA was measured in logMAR (logarithm of the minimum angle of resolution), with 0.00 logMAR corresponding to 20/20 Snellen. A lower logMAR value indicates better visual acuity.
Time Frame: Baseline/Screening (Day 0), Day 1 Postoperative, Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Baseline/Screening (Day 0); Day 1 Postoperative; Month 1 Postoperative; Month 3 Postoperative; Month 6 Postoperative; Month 12 Postoperative: WaveLight Refractive Suite
Arm/Group | Baseline/Screening (Day 0) | Day 1 Postoperative | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 59 | 59 | 59 | 59 | 59
logMAR
  Right eye (OD) | 1.078 (0.4042) | 0.043 (0.1469) | -0.021 (0.1269) | -0.024 (0.1123) | -0.041 (0.0982) | -0.059 (0.1269)
  Left eye (OS) | 1.086 (0.3849) | 0.038 (0.1182) | -0.029 (0.1131) | -0.027 (0.1129) | -0.045 (0.1116) | -0.067 (0.0990)
  Both eyes (OU) | 1.024 (0.4289) | -0.011 (0.1118) | -0.070 (0.0853) | -0.085 (0.0786) | -0.084 (0.0858) | -0.134 (0.0793)

6. Secondary Outcome: Best Corrected Visual Acuity (BCVA)
Description: VA with the subjects's best spectacles or other visual corrective devices, was performed with an ETDRS chart set at a distance of 4 meters. BCVA was measured in logMAR (logarithm of the minimum angle of resolution), with 0.00 logMAR corresponding to 20/20 Snellen. A lower logMAR value indicates better visual acuity.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Baseline/Screening (Day 0) | Day 1 Postoperative | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 59 | 59 | 59 | 59 | 59
logMAR
  Right eye (OD) | -0.046 (0.0855) | -0.028 (0.1097) | -0.064 (0.0953) | -0.072 (0.0877) | -0.091 (0.0810) | -0.103 (0.0880)
  Left eye (OS) | -0.042 (0.0894) | -0.027 (0.0915) | -0.062 (0.0947) | -0.070 (0.0967) | -0.086 (0.0941) | -0.099 (0.0976)
  Both eyes (OU) | -0.063 (0.0814) | -0.051 (0.0973) | -0.096 (0.0907) | -0.099 (0.0863) | -0.111 (0.0870) | -0.148 (0.0837)

7. Secondary Outcome: Manifest Refraction (Sphere)
Description: A series of test lenses in graded powers was used to determine which corrective lenses provided the sharpest, clearest vision. Manifest refraction is measured in diopters. Each eye contributed individually to the analysis.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Eyes
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 59
Number analyzed (Eyes) | 118
Diopters
  Baseline/Screening (Day 0) | -4.254 (2.3340)
  Day 1 Postoperative | -0.347 (0.4174)
  Month 1 Postoperative | -0.186 (0.3304)
  Month 3 Postoperative | -0.153 (0.3049)
  Month 6 Postoperative | -0.167 (0.3253)
  Month 12 Postoperative | -0.165 (0.3190)

8. Secondary Outcome: Manifest Refraction (Cylinder)
Description: as for outcome 7
Time Frame: Baseline/Screening (Day 0), Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: eyes
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 59
Number analyzed (eyes) | 118
Diopters
  Baseline/Screening (Day 0) | -0.95 (0.847)
  Month 1 Postoperative | -0.15 (0.236)
  Month 3 Postoperative | -0.15 (0.251)
  Month 6 Postoperative | -0.16 (0.242)
  Month 12 Postoperative | -0.17 (0.323)

9. Secondary Outcome: Mean Contrast Sensitivity (CS)
Description: Contrast sensitivity (ie, the ability to detect slight changes in luminance before they become indistinguishable) was assessed binocularly with distance manifest correction in place and uncorrected. Contrast sensitivity was assessed at spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd), where 3.0 cpd = A, 6.0 cpd = B, 12.0 cpd = C, and 18.0 cpd = D. Raw scores were log transformed. A higher numeric value represents better contrast sensitivity. Both eyes contributed to the analysis.
Time Frame: Baseline/Screening (Day 0), Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: logCS
Arm/Group | Baseline/Screening (Day 0) | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 59 | 59 | 59 | 59
logCS
  CS A (uncorrected), n=31, 59, 59, 59, 59 | 0.872 (0.5604) | 1.996 (0.1219) | 1.971 (0.1249) | 2.006 (0.1585) | 2.046 (0.1460)
  CS B (uncorrected), n=30, 59, 59, 59, 59 | 0.986 (0.4934) | 2.080 (0.1427) | 2.087 (0.1571) | 2.148 (0.1428) | 2.163 (0.1588)
  CS C (uncorrected), n=28, 59, 58, 59, 58 | 0.687 (0.4789) | 1.802 (0.2096) | 1.802 (0.2009) | 1.833 (0.2259) | 1.866 (0.1727)
  CS D (uncorrected), n=29, 58, 57, 56, 58 | 0.321 (0.5745) | 1.317 (0.2619) | 1.321 (0.2485) | 1.369 (0.2517) | 1.396 (0.2379)
  CS A (corrected), n=59, 59, 59, 59, 59 | 1.970 (0.1576) | 1.993 (0.1310) | 2.003 (0.0967) | 2.025 (0.1424) | 2.076 (0.1126)
  CS B (corrected), n=59, 59, 59, 59, 59 | 2.074 (0.1779) | 2.112 (0.1502) | 2.100 (0.1424) | 2.180 (0.1243) | 2.172 (0.1545)
  CS C (corrected), n=59, 59, 58, 59, 58 | 1.706 (0.2716) | 1.815 (0.2017) | 1.813 (0.1970) | 1.848 (0.2211) | 1.897 (0.1538)
  CS C (corrected), n=57, 58, 57, 56, 58 | 1.262 (0.2657) | 1.338 (0.2713) | 1.332 (0.2491) | 1.388 (0.2501) | 1.422 (0.2292)

10. Secondary Outcome: Corneal Flap Diameter as Assessed by Ocular Coherence Tomography (OCT)
Description: The diameter of the corneal flap was assessed by OCT (ie. an imaging method using light to capture three-dimensional images). Corneal flap is measured in millimeters.
Time Frame: Operation/Surgery (Day 1), Day 1 Postoperative, Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Operation/Surgery (Day 1); Day 1 Postoperative; Month 1 Postoperative; Month 3 Postoperative; Month 6 Postoperative; Month 12 Postoperative: WaveLight Refractive Suite
Arm/Group | Operation/Surgery (Day 1) | Day 1 Postoperative | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 59 | 59 | 59 | 59 | 59
millimeters
  Right eye (OD) | 8.4 (0.25) | 8.4 (0.25) | 8.4 (0.24) | 8.4 (0.25) | 8.4 (0.25) | 8.4 (0.25)
  Left eye (OS) | 8.4 (0.27) | 8.4 (0.27) | 8.4 (0.26) | 8.4 (0.27) | 8.4 (0.27) | 8.4 (0.27)

11. Secondary Outcome: Wavefront Aberrometry
Description: Wavefront aberrations (optical imperfections of the eye that prevent light from focusing perfectly on the retina, resulting in defects in the visual image) were measured using a commercially available system. Higher order aberrations (i.e., spherical aberrations, coma, and trefoil) are defined as optical imperfections which cannot be corrected by any reliable means of present technology.
Time Frame: Operation/Surgery (Day 1), Month 1 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Operation/Surgery (Day 1) | Month 1 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 57 | 59 | 59
micrometers
  Total Higher Order RMS, Right Eye | 0.37 (0.138) | 0.64 (0.517) | 0.60 (0.445) | 0.65 (0.601)
  Total Higher Order RMS, Left eye | 0.40 (0.246) | 0.56 (0.293) | 0.57 (0.318) | 0.58 (0.375)
  Spherical Aberration, Right Eye | 0.0824 (0.13093) | 0.1399 (0.23398) | 0.1646 (0.20307) | 0.1619 (0.19886)
  Spherical Aberration, Left Eye | 0.0851 (0.12651) | 0.1614 (0.20808) | 0.1727 (0.21057) | 0.1954 (0.18350)
  Coma, Right Eye | 0.2059 (0.11420) | 0.3656 (0.34574) | 0.3306 (0.34061) | 0.3416 (0.27229)
  Coma, Left Eye | 0.2040 (0.16540) | 0.2950 (0.16431) | 0.2927 (0.19461) | 0.2858 (0.18065)
  Trefoil, Right Eye | 0.1798 (0.12264) | 0.2316 (0.24752) | 0.2440 (0.22987) | 0.2708 (0.51291)
  Trefoil, Left Eye | 0.2192 (0.18534) | 0.2330 (0.21332) | 0.2400 (0.22751) | 0.2403 (0.20733)

12. Secondary Outcome: Mean Response: "Rate Your Vision, Over the Past 4 Weeks, With NO Glasses or Contact Lenses"
Description: As recorded by the subject on the the Refractive Status and Vision Profile (RSVP), a self-reported questionnaire used to measure vision-related health status in persons with refractive error, on a scale from 0 (completely blind) to 10 (perfect vision).
Time Frame: Baseline/Screening (Day 0), Month 1 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline/Screening (Day 0) | Month 1 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 43 | 59 | 59 | 59
units on a scale | 2.7 (1.42) | 9.0 (1.03) | 9.3 (0.82) | 9.2 (1.06)

13. Secondary Outcome: Percent Response to "Have Always Worn Glasses or Contact Lenses in the Past 4 Weeks"
Description: As recorded by the subject on the the Refractive Status and Vision Profile (RSVP), a self-reported questionnaire used to measure vision-related health status in persons with refractive error.
Time Frame: Baseline/Screening (Day 0), Month 1 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: This analysis population includes all subjects with 1 month post-operative measurements of the primary efficacy endpoint.
Measure: Number; unit: percentage of subjects
Arm/Group | Baseline/Screening (Day 0) | Month 1 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 59 | 59 | 59
percentage of subjects
  No | 67.8 | 100.0 | 100.0 | 100.0
  Yes | 32.2 | 0.0 | 0.0 | 0.0

14. Secondary Outcome: Percent Response by Category: "I Worry About my Vision"
Description: As recorded by the subject on the RSVP questionnaire
Time Frame: Baseline/Screening (Day 0), Month 1 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Baseline/Screening (Day 0) | Month 1 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 59 | 59 | 59
percentage of subjects
  Never | 15.3 | 27.1 | 50.8 | 55.9
  Rarely | 33.9 | 54.2 | 30.5 | 23.7
  Sometimes | 32.2 | 8.5 | 11.9 | 13.6
  Often | 16.9 | 8.5 | 5.1 | 5.1
  Always | 1.7 | 1.7 | 1.7 | 1.7

15. Secondary Outcome: Percent Response by Category: "My Vision is a Concern in my Daily Life"
Description: As recorded by the subject on the RSVP questionnaire
Time Frame: Baseline/Screening (Day 0), Month 1 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Baseline/Screening (Day 0) | Month 1 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 59 | 59 | 59
percentage of subjects
  Never | 3.4 | 27.1 | 44.1 | 50.8
  Rarely | 28.8 | 49.2 | 30.5 | 22.0
  Sometimes | 33.9 | 6.8 | 5.1 | 6.8
  Often | 8.5 | 6.8 | 3.4 | 6.8
  Always | 25.4 | 10.2 | 16.9 | 13.6

16. Secondary Outcome: Percent Response by Category: "Driving at Night"
Description: As recorded by the subject on the RSVP questionnaire, where 0 is "Not applicable", 1 is "No difficulty at all", 2 is "A little difficulty", 3 is "Moderate difficulty", 4 is "Severe difficulty" and 5 is "So much difficulty that I did not do the activity with this alternative".
Time Frame: Baseline/Screening (Day 0), Month 1 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Baseline/Screening (Day 0) | Month 1 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 57 | 59 | 59 | 59
percentage of subjects
  With glasses, 0 | 3.5 | 100.0 | 100.0 | 100.0
  With glasses, 1 | 42.1 | 0.0 | 0.0 | 0.0
  With glasses, 2 | 40.4 | 0.0 | 0.0 | 0.0
  With glasses, 3 | 7.0 | 0.0 | 0.0 | 0.0
  With glasses, 4 | 5.3 | 0.0 | 0.0 | 0.0
  With glasses, 5 | 1.8 | 0.0 | 0.0 | 0.0
  With contact lenses, 0 | 49.1 | 100.0 | 100.0 | 100.0
  With contact lenses, 1 | 35.1 | 0.0 | 0.0 | 0.0
  With contact lenses, 2 | 12.3 | 0.0 | 0.0 | 0.0
  With contact lenses, 3 | 1.8 | 0.0 | 0.0 | 0.0
  With contact lenses, 4 | 0.0 | 0.0 | 0.0 | 0.0
  With contact lenses, 5 | 1.8 | 0.0 | 0.0 | 0.0
  Without glasses/contact lenses, 0 | 33.3 | 6.8 | 5.1 | 5.1
  Without glasses/contact lenses, 1 | 0.0 | 66.1 | 76.3 | 79.7
  Without glasses/contact lenses, 2 | 0.0 | 18.6 | 13.6 | 6.8
  Without glasses/contact lenses, 3 | 1.8 | 6.8 | 5.1 | 3.4
  Without glasses/contact lenses, 4 | 17.5 | 1.7 | 0.0 | 3.4
  Without glasses/contact lenses, 5 | 47.4 | 0.0 | 0.0 | 1.7

17. Secondary Outcome: Corneal Curvature as Measured by Keratometry
Description: Corneal curvature as assessed by a commercially available system and measured in diopters.
Time Frame: Baseline/Screening (Day 0), 1 Month Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: diopter
Arm/Group | Baseline/Screening (Day 0) | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative | Month 12 Postoperative
Number analyzed (Participants) | 59 | 59 | 59 | 59 | 59
diopter
  K1, Right Eye | 43.4 (1.58) | 39.9 (2.42) | 39.9 (2.43) | 40.0 (2.36) | 40.1 (2.34)
  K1, Left Eye | 43.5 (1.74) | 39.8 (2.37) | 39.8 (2.20) | 39.9 (2.31) | 40.0 (2.26)
  K2, Right Eye | 44.6 (1.69) | 40.6 (2.59) | 40.7 (2.52) | 40.8 (2.51) | 40.8 (2.47)
  K2, Left Eye | 44.7 (1.78) | 40.5 (2.49) | 40.5 (2.32) | 40.8 (2.37) | 40.8 (2.35)
  Mean K1 and K2, Right Eye | 44.0 (1.60) | 40.3 (2.47) | 40.3 (2.46) | 40.4 (2.42) | 40.5 (2.39)
  Mean K1 and K2, Left Eye | 44.1 (1.72) | 40.1 (2.42) | 40.2 (2.25) | 40.4 (2.33) | 40.4 (2.30)

18. Secondary Outcome: Flap Creation Time as Documented in the Log Files
Description: The time to create the flap with FS200 Femtosecond Flap Creation System, measured in seconds.
Time Frame: Operation/Surgery (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- FS200 Laser: Femtosecond FS200 laser used during LASIK surgery for corneal flap creation
Arm/Group | FS200 Laser
Number analyzed (Participants) | 59
seconds
  Right eye (OD) | 34.864 (7.3001)
  Left eye (OS) | 33.220 (7.7550)

19. Secondary Outcome: Corneal Topography: Q-value
Description: The Q-value (a measure of corneal asphericity) was assessed using a commercially available system. The Q-values are negative (-1 < Q < 0) for prolate corneas, in which the central curvature is steeper than the peripheral curvature, and positive (Q > 0) for oblate corneas, in which the central curvature is flatter than the peripheral curvature.
Time Frame: Day 1 Postoperative, Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: This analysis population includes all subjects with 1 day post-operation measurements of the corneal topography endpoint. Here, "n" includes all eyes with data.
Measure: Mean (Standard Deviation); unit: unit less
Units Other Than Participants: Eyes
Groups:
- Q-Value: WaveLight Refractive Suite
Arm/Group | Q-Value
Number analyzed (Participants) | 59
Number analyzed (Eyes) | 118
unit less
  Day 1 Postoperative, n=116 | -0.30 (0.661)
  Month 1 Postoperative, n=118 | -0.31 (0.652)
  Month 3 Postoperative, n=118 | -0.06 (0.769)
  Month 6 Postoperative, n=118 | 0.10 (0.752)
  Month 12 Postoperative, n=118 | 0.02 (0.748)

20. Secondary Outcome: Corneal Topography: Anterior Chamber (AC) Volume
Description: The AC volume (a measure of the shallowness of the anterior chamber) was assessed using a commercially available system. The lower the chamber volume, the more shallow the anterior chamber or the chamber angle.
Time Frame: Day 1 Postoperative, Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: millimeters cubed
Units Other Than Participants: Eyes
Groups:
- AC Volume: WaveLight Refractive Suite
Arm/Group | AC Volume
Number analyzed (Participants) | 59
Number analyzed (Eyes) | 118
millimeters cubed
  Day 1 Postoperative, n=116 | 189.98 (30.439)
  Month 1 Postoperative, n=118 | 195.25 (32.134)
  Month 3 Postoperative, n=118 | 192.91 (31.156)
  Month 6 Postoperative, n=118 | 191.92 (32.985)
  Month 12 Postoperative, n=118 | 192.64 (33.382)

21. Secondary Outcome: Corneal Topography: Anterior Chamber (AC) Depth
Description: The AC depth (axial distance between the anterior surface of the cornea and the anterior surface of the lens) was assessed using a commercially available system. A higher value represents a longer distance.
Time Frame: Day 1 Postoperative, Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Groups:
- AC Depth: WaveLight Refractive Suite
Arm/Group | AC Depth
Number analyzed (Participants) | 59
Number analyzed (Eyes) | 118
millimeters
  Day 1 Postoperative, n=116 | 3.43 (0.370)
  Month 1 Postoperative, n=117 | 3.43 (0.349)
  Month 3 Postoperative, n=118 | 3.38 (0.352)
  Month 6 Postoperative, n=118 | 3.18 (0.272)
  Month 12 Postoperative, n=118 | 3.16 (0.276)

22. Secondary Outcome: Corneal Topography: Angles
Description: The angles (angular measurement of the space between the iris and the lens) were assessed using a commercially available system. The higher the value, the bigger the space.
Time Frame: Day 1 Postoperative, Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative, Month 12 Postoperative
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Eyes
Groups:
- Angles: WaveLight Refractive Suite
Arm/Group | Angles
Number analyzed (Participants) | 59
Number analyzed (Eyes) | 118
degrees
  Day 1 Postoperative, n=116 | 41.07 (6.612)
  Month 1 Postoperative, n=118 | 40.63 (6.155)
  Month 3 Postoperative, n=118 | 41.09 (6.155)
  Month 6 Postoperative, n=118 | 40.81 (6.141)
  Month 12 Postoperative, n=118 | 40.74 (6.133)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 12 months). This reporting group includes all enrolled subjects who underwent LASIK surgery.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device.
Arm/Group | WaveLight Refractive Suite
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.